CLINICAL TRIAL: NCT01262547
Title: A Randomized Controlled Pilot Study to Examine the Use of Micrografting, Using a Novel Grafting Technique for the Repigmentation of Vitiligo
Brief Title: A New Micrografting Technique for Vitiligo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study sponsor was acquired by a company that focuses on chronic wounds.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Momelan Technologies (Industry)
Responsible Party: Principal Investigator, Alexandra Kimball, Director, Clinical Unit for Research Trials in Skin, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-p-001784
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Dermabrasion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dermabrasion-Micrografting (Experimental): Dermabrasion-Micrografting
  Interventions: Device: Dermabrasion-Micrografting
- Dermabrasion alone (Active Comparator): Dermabrasion alone
  Interventions: Procedure: Dermabrasion
- Control (No Intervention): Control

INTERVENTIONS:
Device: Dermabrasion-Micrografting — Several small pieces of skin, each measuring 1.75 mm in diameter will be harvested from a normal pigmented area using a commercially available suction blister device. This will be attached to a sterile elastomeric substrate and then placed on a recipient area prepared by epidermal dermabrasion (removal of the epidermis).
  Arms: Dermabrasion-Micrografting
Procedure: Dermabrasion — Only dermabrasion (removal of epidermis) alone will be done at baseline.
  Arms: Dermabrasion alone

SUMMARY:
This study evaluates micrografting using a harvesting and grafting process that has been designed by Momelan Technologies. The overall concept is to harvest several small pieces of skin, each measuring about 1.75 mm in diameter from a normal pigmented area using a commercially available suction blister device, adhere them to a sterile elastomeric substrate and is then place it on a recipient area prepared by epidermal dermabrasion (removal of the epidermis).

DETAILED DESCRIPTION:
Participants with vitiligo patches undergo removal of the epidermis of the affected vitiligo skin with dermabrasion. Several small pieces of pigmented skin (1.75mm) from the patient are taken from another area with the use of a suction blister device. The harvested pigmented skin is adhered to a sterile elastomeric substrate and placed on the previously dermabraded affected area.

Originally the primary outcome was percentage of change in pigmentation with UV photos at 10 weeks in sites undergoing grafts compared to control sites. However, because we were unable to take UV photos, we had to revise our primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 to 80 years old
* Have a diagnosis of stable vitiligo as defined by Vitiligo Disease Activity Score of 0 or 1
* Has 3 comparable vitiliginous areas of trunk or extremities (excluding hands) each measuring at least 3cm×3cm in size, with at least 80% of depigmentation, and anticipated equal sun exposure.
* Have not used any topical therapy to patches or Ultraviolet light therapy for at least 2 weeks (subjects may restart phototherapy at week 10 if desired)
* Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form
* Agree to follow and undergo all study-related procedures

Exclusion Criteria:

* Female patients who are breastfeeding, pregnant, or planning to become pregnant
* Patients with a history of hypertrophic scaring or keloids and psoriasis
* Subjects on any dose of coumadin, warfarin, Plavix or at least 325 mg aspirin.
* Concurrent use of immunosuppressive medications such as oral steroids, tacrolimus and other cytotoxic reagents within 2 weeks of grafting)
* Subject who received topical therapy or UV light ( phototherapy)in last 2 weeks
* Patients with a positive HIV status
* Patients withDiabetes Mellitus with a hemoglobin A1C of more than 8.
* Subjects with dermatologic conditions that may Koebnerize such as psoriasis and lichen planus.
* Participation in another interventional study with potential exposure to an investigational drug within past 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B Kimball, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mgh Curtis, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Vitiligo: Three subjects with vitiligo were recruited for the study. All subjects had three test sites that were studied. One site received dermabrasion and micrografting, one site received dermabrasion alone and one site was not treated and served as the control.
Period: Overall Study
Arm/Group | Patients With Vitiligo
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Dermabrasion-Micrografting, Dermabrasion and Control
  Dermabrasion-Micrografting: Several small pieces of skin, each measuring 1.75 mm in diameter will be harvested from a normal pigmented area using a commercially available suction blister device. This will be attached to a sterile elastomeric substrate and then placed on a recipient area prepared by epidermal dermabrasion (removal of the epidermis).
  Dermabrasion: Only dermabrasion (removal of epidermis) alone will be done at baseline.
  Control: Untreated depigmented area
Arm/Group | All Study Participants
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 47 [43 to 53]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Target VASI Score From Baseline to Week 24.
Description: Target Vitiligo Area Scoring Index (VASI) consists of a 7-point scale ranging from 0 (no change in depigmentation) to 6 (complete repigmentation).
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Control: Target sites did not receive any treatment
Arm/Group | Dermabrasion-Micrografting | Dermabrasion Alone | Control
Number analyzed (Participants) | 3 | 3 | 3
units on a scale | 0.33 [0 to 1] | 0.33 [0 to 1] | 0 [0 to 0]

2. Secondary Outcome: Incidence of Adverse Effects, Including Increased Activity of Vitiligo
Time Frame: 24 weeks
Measure: Number; unit: participants reporting redness
Arm/Group | Dermabrasion-Micrografting | Dermabrasion Alone | Control
Number analyzed (Participants) | 3 | 3 | 3
participants reporting redness | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: 24 Weeks
Groups:
- Control: Control
  Depigmented areas that did not receive any treatment.
Arm/Group | Dermabrasion-Micrografting | Dermabrasion Alone | Control
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dermabrasion-Micrografting (N=3) | Dermabrasion Alone (N=3) | Control (N=3)
Mild Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0
Moderate Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0

LIMITATIONS AND CAVEATS:
Early termination of study leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No